CLINICAL TRIAL: NCT04281056
Title: Impact of Complete Tooth Loss and Denture on Oral Sensory Abilities and Food Preference
Brief Title: Impact of Tooth Loss and Denture on Oral Senses and Food Preferences
Acronym: AlimaPAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP190340
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Tooth-loss
Keywords: Teeth loss; edentulousness; denture; tast; trigeminal senses; oral sensory ability
MeSH Terms: conditions — Anodontia | interventions — Tooth Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Tooth removal (Experimental): Tooth removal and their replacement by means of a denture Teeth have been removed and replaced by means of dentures for at least one year
  Interventions: Procedure: Tooth removal and their replacement by means of a denture

INTERVENTIONS:
Procedure: Tooth removal and their replacement by means of a denture — Teeth have been removed and replaced by means of dentures for at least one year
  Arms: Tooth removal

SUMMARY:
Tooth loss impacts taste abilities and food intake. Present study aims at pertaining the impact of teeth loss and the replacement by means of complete denture on taste and trigeminal abilities, and on food preferences, and taste appetence.

DETAILED DESCRIPTION:
Two groups of participants will be included. Participants wearing complete denture for at least one year (n=20) and their matched controls for age, sex, tobacco, and saliva secretion (n=20). Their oral sensory abilities of participants will be assessed including taste (electrogustometric thresholds, chemical taste identification ability) and trigeminal quantitative sensory testing. Food preferences and selectivity (Maitre et al., 2014) and taste appetence (Deglaire et al., 2012) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

Study Group : being completely edentulous and wearing denture for at least one year, wearing denture during meals, with clean and stable dentures. Controls:

controls Group : dentate subjects (25 teeth at leas, non endodontically treated) with molars in Angle's Class I occlusion, having no functional disturbance of mastication and not undergoing dental treatment at the time of the recording. Matched with subjects of the study group for age, sex, tabacco consumption, and saliva flow rate.

Exclusion Criteria:

* Aged under 18 or over 80 Y,
* not consenting to participate
* suffering from dental
* periodontal or gum pain for the last month.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
taste detection thresholds | up to 30 days
  Using an Electrogustometer

SECONDARY OUTCOMES:
Chemical taste identification ability | up to 30 days
  Using taste strips (Burghard)
Quantitative sensory testing | up to 30 days
  Using an algometer, von frey filament, a thermode.
Food preferences and selectivity | up to 30 days
  Questionnaire food selectyivity and preference (Maitre et al., 2014)
Taste appetence | up to 30 days
  Questionnaire PrefQuest (Deglaire et al., 2012)

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Braud, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service odontologie Hôpital Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No